CLINICAL TRIAL: NCT06775392
Title: Comparative Evaluation of Bromelain-Quercetin Gel With Chlorhexidine Gel as Subgingival Local Drug Delivery Following Scaling and Root Planing In Stage I /II and Grade B Periodontitis - Randomized Control Clinical Trail
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCDSHEC/IP/2023/V1/P4a
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-1-SRP alone (Active Comparator): control group is treated with SRP alone
  Interventions: Procedure: SRP
- Group-2-2%bromelain-quercetin gel (Experimental): test group treated with 2%bromelain-quercetin gel
  Interventions: Drug: bromelain-quercetin gel
- Group-3-0.2% chlorhexidine gel (Active Comparator): test group treated with chlorhexidine gel
  Interventions: Drug: chlorhexidine gel

INTERVENTIONS:
Drug: bromelain-quercetin gel — bromelain-quercetin gel is prepared from capsules in laboratory
  Arms: Group-2-2%bromelain-quercetin gel
Drug: chlorhexidine gel — chlorhexidine gel is prepared in laboratory
  Arms: Group-3-0.2% chlorhexidine gel
Procedure: SRP — Scaling and root planing was done with ultra sonic and hand scaling
  Arms: Group-1-SRP alone

SUMMARY:
Comparative Evaluation of Bromelain-Quercetin Gel With Chlorhexidine Gel as Subgingival Local Drug Delivery Following Scaling and Root Planing In Stage I /II and Grade B Periodontitis - Randomized Control Clinical Trail

DETAILED DESCRIPTION:
: Periodontitis is a biofilm associated disease that induces an irreversible inflammatory state that leads to the destruction of the supporting structure of the teeth. Management of periodontal disease is through thorough removal of biofilm which is pivotal for having better oral health. Scaling and root planning (SRP) is fundamental treatment for periodontitis. Years of documented research have established that chlorhexidine digluconate (CHX), gold standard of chemical plaque control agent is safe stable and effective in preventing and controlling plaque formation. Bromelain is an extract derived from Ananas comosus (popularly known as pineapple), contains proteinases that exhibits anti-inflammatory properties, antibacterial effect against periodontopathogens. Bromelain gel has shown to have chemicomechanical method of caries removal. Quercetin present in guava have excellent antibacterial actions against periodontal pathogens, Aggregatibacter actinomycetemcomitans (Aa), Porphyromonas gingivalis (Pg), Prevotella intermedia (Pi) and Fusobacterium nucleatum (Fn). 2% Quercetin has shown to be advantageous for subgingival application after scaling and rootplaning. Bromelain-Quercetin gel has shown adjunctive effect for treatment in covid-19 patients. As there is less literature in this combination, we intend to study its effects. Individually bromelain and quercetin have been studied for treatment in oral cavity as gel form. This study will be first of its kind to check the efficacy of 2% bromelain-quercetin gel and to compare its effects with 0.2% Chlorhexidine in stage I/II and grade B periodontits.

ELIGIBILITY:
Inclusion Criteria:

* Patient with have chronic periodontitis in the age group between 30-50 years.
* Patients having ≥20 teeth.

  -.Patients with radiographic evidence of bone loss in atleast two teeth.
* Patients who are systematically healthy.
* Patients with localized pockets with probing depth of ≤ 5mm.
* Patients who are cooperative and able to attend the hospital for regular follow-up.

Exclusion Criteria:

* Patients who have received any surgical or nonsurgical therapy during past 6months
* Pregnant or lactating females.
* Use of systemic antibiotics in the past 6 months.
* Patient who are not willing to give a written informed consent

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
PROBING POCKET DEPTH | 21DAYS
  measured using a UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA
CLINICAL ATTACHMENT LEVEL | 21DAYS
  (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Plaque Index | 21DAYS
  measured on the tooth surface using a probe
Gingival index | 21DAYS
  measured on the tooth surface using a probe
Modified Sulcus Bleeding Index | 21days
  measured on the tooth surface using a probe

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. NALLAGATLA VAMSI VENKATA KRISHNA SAI, Bengaluru, Karnataka, India